CLINICAL TRIAL: NCT06704841
Title: Effect of Music and Mindfulness Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Teresa Lesiuk, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20241057
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music in combination with mindfulness group (Experimental): Participants in this group will receive music in combination with mindfulness group for up to two weeks.
  Interventions: Behavioral: Music in combination with mindfulness

INTERVENTIONS:
Behavioral: Music in combination with mindfulness — Participants will attend two in-person sessions per week over two consecutive weeks. Each session will be up to one hour in duration. During each session, participants will engage in a 20-minute guided meditation while listening to instrumental music.

SUMMARY:
The purpose of the study is to explore the effect of music and mindfulness meditation on anxiety and mindful interoception in undergraduate music students.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be undergraduate college students majoring in a music degree.
* Participants must self-report feeling general anxiety at a level of 7/10 recently.
* Participants must be proficient English-readers and -speakers and be full-time enrolled students.
* Students of any gender and race/ethnic group may be included.
* Participants must be novice meditators, having fewer than 10 total meditation experiences.
* Students of any year will be accepted if they are considered undergraduate students by the university.

Exclusion Criteria:

* Self-reporting feeling general anxiety below a 7/10 recently.
* Having more than 10 total meditation experiences.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Change in State-Anxiety Inventory-5 questionnaire | Baseline, up to 1 hour post intervention
  The State-Anxiety Inventory-5 each consists of 5 items. The scale items are scored on a 4-point Likert scale of 1 to 4 (1= Not at all, 2= Somewhat, 3= Moderately so, 4= Very much so). Higher scores indicate greater anxiety.

SECONDARY OUTCOMES:
Change in Mindfulness Interoception measured by Likert scale | Baseline, 2 weeks
  The scale items are scored on a 4-point Likert scale of 1 to 4 (1= Not at all, 2= Somewhat, 3= Moderately so, 4= Very much so). A higher score suggests higher mindful interoception skills.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Lesiuk, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No